CLINICAL TRIAL: NCT05950724
Title: RENAL: Randomized Clinical Trial of TNF-alpha Inhibitor for Improving Renal Dysfunction and Primary Graft Dysfunction After Lung Transplant
Brief Title: RENAL: TNF-alpha Inhibitor for Improving Renal Dysfunction and Primary Graft Dysfunction After Lung Transplant
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Chitaru Kurihara, Instructor of Surgery, Feinberg School of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU00218926
Record Dates: First submitted 2023-07-03; First posted 2023-07-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lung Transplant; Complications
MeSH Terms: interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Etanercept (Experimental): Participants receive one dose (25mg) Etanercept via subcutaneous injection just prior to lung transplant. Following transplant, participants receive standard lung transplant care.
  Interventions: Drug: Etanercept Injection [Enbrel]
- Control (No Intervention): Participants receive standard lung transplant care.

INTERVENTIONS:
Drug: Etanercept Injection [Enbrel] — 25 mg subcutaneous injection
  Arms: Etanercept

SUMMARY:
The purpose of this study is to assess whether TNFa antibody use before lung transplant can prevent kidney injury after lung transplant.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written consent who undergo a lung transplant will be randomized in a 1:1 ratio to either the treatment or control group. Patients randomized to the treatment group will receive one dose of the study drug, Etanercept, via subcutaneous injection just prior to the lung transplant. Patients randomized to the control group will not receive Etanercept. Both groups will receive standard lung transplant care after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Planning to undergo transplantation of the lung at Northwestern Memorial Hospital.
* Willing and able to read, understand, and be capable of giving informed consent.

Exclusion Criteria:

* Previous or current use of TNFa antibody.
* Positive virtual or retrospective crossmatch or highly sensitized (pRA > 30%) recipients.
* Any condition that, in the opinion of the attending physician, would place the patient at undue risk by participating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of kidney dysfunction immediately after lung transplant | Immediately after lung transplant
  Measured by serum creatinine blood tests
Occurrence of kidney dysfunction post-operatively within 1 week after lung transplant | Within 1-7 days after lung transplant
  Measured by serum creatinine blood tests
Occurrence of kidney dysfunction post-operatively within 1 month after lung transplant | Up to 30 days after lung transplant
  Measured by serum creatinine blood tests

SECONDARY OUTCOMES:
Occurrence of primary graft dysfunction | Within 3 days post-transplant
  Measured by arterial blood gas (ABG) blood tests and chest X-rays
Length of intensive care unit (ICU) stay | Through study completion, an average of 1 year
  Measured by number of days in the ICU post-transplant
Length of ventilator use | Through study completion, an average of 1 year
  Measured by number of days on a ventilator post-transplant
Survival | 30 days, 90 days, and one year survival post-transplant
  Alive or dead post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Chitaru Kurihara, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnold CM, Bailey DA, Faulkner RA, McKay HA, McCulloch RG. The effect of water fluoridation on the bone mineral density of young women. Can J Public Health. 1997 Nov-Dec;88(6):388-91. doi: 10.1007/BF03403912. PMID 9458565
- [Background] Wajda-Pokrontka M, Nadziakiewicz P, Krauchuk A, Ochman M, Zawadzki F, Przybylowski P. Influence of Fluid Therapy on Kidney Function in the Early Postoperative Period After Lung Transplantation. Transplant Proc. 2022 May;54(4):1115-1119. doi: 10.1016/j.transproceed.2022.02.021. Epub 2022 Apr 13. PMID 35428509
- [Background] Gerriets V, Goyal A, Khaddour K. Tumor Necrosis Factor Inhibitors. 2023 Jul 3. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482425/ PMID 29494032
- [Background] Meroni PL, Valentini G, Ayala F, Cattaneo A, Valesini G. New strategies to address the pharmacodynamics and pharmacokinetics of tumor necrosis factor (TNF) inhibitors: A systematic analysis. Autoimmun Rev. 2015 Sep;14(9):812-29. doi: 10.1016/j.autrev.2015.05.001. Epub 2015 May 15. PMID 25985765
- [Background] Komaki Y, Yamada A, Komaki F, Kudaravalli P, Micic D, Ido A, Sakuraba A. Efficacy, safety and pharmacokinetics of biosimilars of anti-tumor necrosis factor-alpha agents in rheumatic diseases; A systematic review and meta-analysis. J Autoimmun. 2017 May;79:4-16. doi: 10.1016/j.jaut.2017.02.003. Epub 2017 Feb 13. PMID 28209290
- [Background] Rubbert-Roth A, Atzeni F, Masala IF, Caporali R, Montecucco C, Sarzi-Puttini P. TNF inhibitors in rheumatoid arthritis and spondyloarthritis: Are they the same? Autoimmun Rev. 2018 Jan;17(1):24-28. doi: 10.1016/j.autrev.2017.11.005. Epub 2017 Nov 3. PMID 29108829
- [Background] Haraoui B. Differentiating the efficacy of the tumor necrosis factor inhibitors. Semin Arthritis Rheum. 2005 Apr;34(5 Suppl1):7-11. doi: 10.1016/j.semarthrit.2005.01.003. PMID 15852248
- [Background] Gottlieb AB. Tumor necrosis factor blockade: mechanism of action. J Investig Dermatol Symp Proc. 2007 May;12(1):1-4. doi: 10.1038/sj.jidsymp.5650029. PMID 17502861
- [Background] Roach DR, Bean AG, Demangel C, France MP, Briscoe H, Britton WJ. TNF regulates chemokine induction essential for cell recruitment, granuloma formation, and clearance of mycobacterial infection. J Immunol. 2002 May 1;168(9):4620-7. doi: 10.4049/jimmunol.168.9.4620. PMID 11971010
- [Background] Mocci G, Marzo M, Papa A, Armuzzi A, Guidi L. Dermatological adverse reactions during anti-TNF treatments: focus on inflammatory bowel disease. J Crohns Colitis. 2013 Nov;7(10):769-79. doi: 10.1016/j.crohns.2013.01.009. Epub 2013 Mar 1. PMID 23453887
- [Background] Carcinoma of hypopharynx and cervical oesophagus. Br Med J. 1967 Jun 17;2(5554):718. doi: 10.1136/bmj.2.5554.718. No abstract available. PMID 6025976
- [Background] Tsuhako S. [Beginning course of English medical terminology based on analytical method]. Sogo Kango. 1994 May;29(2):91-4. No abstract available. Japanese. PMID 8026186
- [Background] Puffer LB Jr. Legal problems of the intensive care unit. Med Clin North Am. 1971 Sep;55(5):1365-74. doi: 10.1016/s0025-7125(16)32473-7. No abstract available. PMID 5568853
- [Background] Horn SD. Overview of current models for prospective payment. ANA Publ. 1984 Apr;(G-164):24-35. No abstract available. PMID 6428256
- [Background] Grivennikov SI, Tumanov AV, Liepinsh DJ, Kruglov AA, Marakusha BI, Shakhov AN, Murakami T, Drutskaya LN, Forster I, Clausen BE, Tessarollo L, Ryffel B, Kuprash DV, Nedospasov SA. Distinct and nonredundant in vivo functions of TNF produced by t cells and macrophages/neutrophils: protective and deleterious effects. Immunity. 2005 Jan;22(1):93-104. doi: 10.1016/j.immuni.2004.11.016. PMID 15664162